CLINICAL TRIAL: NCT00371345
Title: Phase II Study of Dasatinib (BMS-354825) for Advanced Estrogen/Progesterone Receptor-Positive or Her2/Neu-Positive Breast Cancer
Brief Title: Study of Dasatinib (BMS-354825) in Patients With Advanced Estrogen/Progesterone Receptor-positive (ER+/PR+) or Her2/Neu-positive (Her2/Neu+)Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-088
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Results first posted 2010-11-05 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer; Metastasis
Keywords: Recurrent, locally-advanced, or metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental): Participants with either a Human epidermal growth factor (Her2/neu)-amplified tumor type or ER and/or PgR positive tumor types received oral dasatinib twice daily (BID).
  Interventions: Drug: Dasatinib; Drug: Dasatinib 100 mg

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 70 mg, twice daily, as long as the participant benefits (average <6 months)
  Other Names: Sprycel; BMS-354825
Drug: Dasatinib 100 mg — Tablets, Oral, 100mg, twice daily, as long as the participant benefits (average <6 months)
  Other Names: Sprycel; BMS-354825

SUMMARY:
This study will determine whether the investigational drug dasatinib is effective in treatment of women with progressive advanced ER+/PR+ or Her2/neu+ breast cancer

ELIGIBILITY:
Inclusion Criteria:

* females, 18 or older
* recurrent, locally advanced, or metastatic breast cancer with expression of ER/PR receptor and/or overexpression of Her2/neu
* paraffin-embedded tissue block must be available
* measurable disease
* prior chemotherapy with an anthracycline and/or a taxane (neoadjuvant, adjuvant, or metastatic setting)
* 0, 1 or 2 chemotherapies in the metastatic setting
* adequate organ function

Exclusion Criteria:

* Metastatic disease confined to bone only
* Symptomatic central nervous system (CNS) metastasis
* Concurrent medical condition which may increase the risk of toxicity
* Unable to take oral medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (7):
  - Ucsf-Comprehensive Cancer Center, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Dana-Farber Cancer Inst, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University Of Texas Md Anderson Cancer Ctr, Houston, Texas
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Haedo, Buenos Aires
- Local Institution, Brussels, Belgium
- France (4):
  - Local Institution, Dijon
  - Local Institution, Paris
  - Local Institution, Saint-Herblain
  - Local Institution, Toulouse
- Local Institution, Modena, Italy
- Peru (2):
  - Local Institution, Arequipa, Arequipa
  - Local Institution, Lima, Lima Province
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Lleida
  - Local Institution, Madrid

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 92 participants were enrolled in the study. Twenty-two participants did not enter the treatment phase, 13 because they did not meet entry criteria and 9 for other reasons. The 70 participants treated in the single-arm were stratified by tumor type into Her2-amplified and ER/PgR positive tumors.
Groups:
- Her2/Neu-amplified Tumor Type: Participants with a Human epidermal growth factor (Her2/neu)-amplified tumor type (defined as 3+ by immunohistochemistry [IHC] or positive by fluorescent or chromogenic in situ hybridization [FISH or CISH] regardless of estrogen receptor [ER]/progesterone receptor [PgR] status) received orally 100 mg of dasatinib twice daily (BID) for a total daily dose (TDD) of 200 mg.
- ER and/or PgR Positive Tumor Type: Participants with ER and/or PgR positive tumor types (defined as >10% of cells positive by IHC [unless Her2/neu-amplified]) received orally 100 mg of dasatinib twice daily (BID) for a total daily dose (TDD) of 200 mg.
Period: Overall Study
Arm/Group | Her2/Neu-amplified Tumor Type | ER and/or PgR Positive Tumor Type
Started | 24 | 46
Completed | 0 | 0
Not Completed | 24 | 46
Not completed — Disease Progression | 21 | 35
Not completed — Study Drug Toxicity | 1 | 7
Not completed — Adverse event(AE Unrelated to Study Drug | 1 | 2
Not completed — Participant Request | 1 | 1
Not completed — Participant Withdrew Consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Her2/Neu-amplified Tumor Type | ER and/or PgR Positive Tumor Type | Total
Number analyzed (Participants) | 24 | 46 | 70
Age Continuous [Mean (Full Range); unit: years] | 52.2 [32 to 68] | 54.3 [33 to 70] | 53.6 [32 to 70]
Age, Customized [Number; unit: participants]
  <=50 years | 8 | 16 | 24
  >=50 years | 16 | 30 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 46 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 9 | 2 | 11
  United States | 10 | 17 | 27
  Argentina | 0 | 6 | 6
  Spain | 4 | 8 | 12
  Belgium | 1 | 10 | 11
  Peru | 0 | 1 | 1
  Italy | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Tumor response was assessed according RECIST criteria: PR=at least 30% reduction in the sum of the LD of all target lesions in reference to the baseline sum LD, CR=Disappearance of all non-target lesions. Objective tumor response was defined as a PR or CR.
Time Frame: From day of first treatment through Week 25 or at time of discontinuation from study treatment.
Population: Evaluable population (n=69): Response Evaluable=treated participants with ≥1 measurable lesion at baseline and ≥1 on-study tumor assessment. One participant was not evaluable (no on-study tumor assessment for other reason).
Measure: Number; unit: participants
Groups:
- Her2/Neu-amplified Tumor, 70 mg Twice Daily (BID) Dasatinib: Participants with a Human epidermal growth factor (Her2/neu)-amplified tumor type (defined as 3+ by immunohistochemistry [IHC] or positive by fluorescent or chromogenic in situ hybridization [FISH or CISH] regardless of estrogen receptor [ER]/progesterone receptor [PgR] status) received orally 70 mg of dasatinib twice daily (BID) for a total daily dose (TDD) of 140 mg.
- Her2/Neu-amplified Tumor, 100 mg BID: Participants with a Human epidermal growth factor (Her2/neu)-amplified tumor type (defined as 3+ by immunohistochemistry [IHC] or positive by fluorescent or chromogenic in situ hybridization [FISH or CISH] regardless of estrogen receptor [ER]/progesterone receptor [PgR] status) received orally 100 mg of dasatinib twice daily (BID) for a total daily dose (TDD) of 200 mg.
- ER and/or PgR Positive Tumor, 70 mg BID Dasatinib: Participants with ER and/or PgR positive tumor types (defined as >10% of cells positive by IHC [unless Her2/neu-amplified]) received orally 70 mg of dasatinib twice daily (BID) for a total daily dose (TDD) of 140 mg.
- ER and/or PgR Positive Tumor, 100 mg BID Dasatinib: Participants with ER and/or PgR positive tumor types (defined as >10% of cells positive by IHC [unless Her2/neu-amplified]) received orally 100 mg of dasatinib twice daily (BID) for a total daily dose (TDD) of 200 mg.
Arm/Group | Her2/Neu-amplified Tumor, 70 mg Twice Daily (BID) Dasatinib | Her2/Neu-amplified Tumor, 100 mg BID | ER and/or PgR Positive Tumor, 70 mg BID Dasatinib | ER and/or PgR Positive Tumor, 100 mg BID Dasatinib
Number analyzed (Participants) | 15 | 9 | 31 | 14
participants | 0 | 1 | 1 | 1

2. Primary Outcome: Percentage of Participants With Objective Response
Description: Tumor response was assessed according RECIST criteria: PR=at least 30% reduction in the sum of the LD of all target lesions in reference to the baseline sum LD, CR=Disappearance of all non-target lesions. Percentage of participants with objective tumor response was determined by the number of participants with PR or CR divided by the total number of response-evaluable participants.
Time Frame: From day of first treatment through Week 25 or at time of discontinuation from study treatment
Population: Evaluable population (n=69): Response Evaluable=treated participants with ≥1 measurable lesion at baseline and ≥1 on-study tumor assessment; Non-responders=treated participants with no on-study tumor response assessment due to rapid disease progression/dasatinib toxicity. One participant was not evaluable (no on-study tumor assessment).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Her2/Neu-amplified Tumor, 100 mg BID Dasatinib: Participants with a Human epidermal growth factor (Her2/neu)-amplified tumor type (defined as 3+ by immunohistochemistry [IHC] or positive by fluorescent or chromogenic in situ hybridization [FISH or CISH] regardless of estrogen receptor [ER]/progesterone receptor [PgR] status) received orally 100 mg of dasatinib twice daily (BID) for a total daily dose (TDD) of 200 mg.
- All Response-evaluable Participants: Evaluable population (n=69): Response Evaluable=treated participants with ≥1 measurable lesion at baseline and ≥1 on-study tumor assessment; Non-responders=treated participants with no on-study tumor response assessment due to rapid disease progression/dasatinib toxicity. One participant was not evaluable (no on-study tumor assessment).
Arm/Group | Her2/Neu-amplified Tumor, 70 mg Twice Daily (BID) Dasatinib | Her2/Neu-amplified Tumor, 100 mg BID Dasatinib | ER and/or PgR Positive Tumor, 70 mg BID Dasatinib | ER and/or PgR Positive Tumor, 100 mg BID Dasatinib | All Response-evaluable Participants
Number analyzed (Participants) | 15 | 9 | 31 | 14 | 69
percentage of participants | 0 [0 to 0] | 11.11 [0.28 to 48.25] | 3.23 [0.08 to 16.70] | 7.14 [0.18 to 33.87] | 4.35 [0.91 to 12.18]

3. Secondary Outcome: Number of Response-evaluable Participants With Disease Control (DCR)
Description: Disease control was defined in response-evaluable participants as having a best response of CR or PR (or uPR), or SD at/after 16 Weeks.
Time Frame: From day of first treatment through Week 25 or at time of discontinuation from study treatment.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Her2/Neu-amplified Tumor, 70 mg Twice Daily (BID) Dasatinib | Her2/Neu-amplified Tumor, 100 mg BID Dasatinib | ER and/or PgR Positive Tumor, 70 mg BID Dasatinib | ER and/or PgR Positive Tumor, 100 mg BID Dasatinib
Number analyzed (Participants) | 1 | 1 | 5 | 2
participants
  Participants with CR | 0 | 0 | 0 | 0
  Participants with unconfirmed PR (uCR) | 0 | 0 | 1 | 0
  Participants with PR | 0 | 1 | 1 | 1
  Participants with SD ≥16 weeks | 1 | 0 | 3 | 1
  Total Participants with DCR | 1 | 1 | 5 | 2

4. Secondary Outcome: Percentage of Response-evaluable Participants With Disease Control (DCR)
Description: Disease control was defined in response-evaluable participants as having a best response of objective response (CR or PR) or SD at/after 16 Weeks.
Time Frame: From day of first treatment through Week 25 or at time of discontinuation from study treatment.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Her2/Neu-amplified Tumor, 70 mg Twice Daily (BID) Dasatinib | Her2/Neu-amplified Tumor, 100 mg BID Dasatinib | ER and/or PgR Positive Tumor, 70 mg BID Dasatinib | ER and/or PgR Positive Tumor, 100 mg BID Dasatinib
Number analyzed (Participants) | 15 | 9 | 31 | 14
percentage of participants | 6.67 [0.17 to 31.95] | 11.11 [0.28 to 48.25] | 16.13 [5.54 to 33.73] | 14.29 [1.78 to 42.81]

5. Secondary Outcome: Number of Participants Who Progressed
Description: PFS was defined as time from first dosing date until the first date that Progressive Disease (PD) was observed.
Time Frame: From Baseline (Week 0) to time of PD or discontinuation of last participant from study treatment (Week 45)
Population: All-Treated subjects: All subjects who received at least one dose of dasatinib. The longest on-study observation for a participant was 45 weeks.
Measure: Number; unit: participants
Groups:
- Her2/Neu-amplified Tumor: Participants with a Human epidermal growth factor (Her2/neu)-amplified tumor type (defined as 3+ by immunohistochemistry [IHC] or positive by fluorescent or chromogenic in situ hybridization [FISH or CISH] regardless of estrogen receptor [ER]/progesterone receptor [PgR] status) received orally dasatinib twice daily (BID).
- ER and/or PgR Positive Tumor: Participants with ER and/or PgR positive tumor types (defined as >10% of cells positive by IHC [unless Her2/neu-amplified]) received orally dasatinib twice daily (BID).
- All Participants: Dasatinib was administered orally at 70 mg BID (TDD=140 mg) or 100 mg BID (TDD=200 mg).
Arm/Group | Her2/Neu-amplified Tumor | ER and/or PgR Positive Tumor | All Participants
Number analyzed (Participants) | 24 | 46 | 70
participants | 22 | 39 | 61

6. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS was defined as time from first dosing date until the first date that PD was observed. The distribution of PFS was estimated using the Kaplan-Meier product limit method. A two-sided 95% confidence interval (Brookmeyer and Crowley method) for the median PFS was computed.
Time Frame: From Baseline (Week 0) to time of PD or discontinuation of last participant from study treatment (Week 45)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Her2/Neu-amplified Tumor | ER and/or PgR Positive Tumor
Number analyzed (Participants) | 24 | 46
weeks | 8.1 [7.1 to 9.3] | 8.1 [7.7 to 8.7]

7. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS) at Weeks 9, 17, and 25
Description: PFS was defined as time from first dosing date until the first date that progressive disease (PD) was observed.
Time Frame: At Weeks 9, 17, and 25
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Her2/Neu-amplified Tumor, 70 mg Twice Daily (BID) Dasatinib | Her2/Neu-amplified Tumor, 100 mg BID Dasatinib | ER and/or PgR Positive Tumor, 70 mg BID Dasatinib | ER and/or PgR Positive Tumor, 100 mg BID Dasatinib
Number analyzed (Participants) | 15 | 9 | 32 | 14
percentage of participants
  Week 9 | 21 | 50 | 32 | 33
  Week 17 | 7 | 25 | 18 | 25
  Week 25 | 0 | 13 | 7 | 17

8. Secondary Outcome: Duration Of Objective Response
Description: Duration of objective response was defined as the time (in weeks) between the first date that criteria for CR or PR were met and the first date that progressive disease (PD) or clinical progressive disease (cPD) was observed. Date of death was used as PD date for participants who died before reporting PD. Participants who neither progressed nor died were censored at the date of their last tumor assessment.
Time Frame: the time (in weeks) between the first date that criteria for PR were met and the first date that PD or cPD was observed
Population: Of 69 response-evaluable participants, three had an objective response of PR.
Measure: Number; unit: weeks
Groups:
- Participant CA180088-18-88009, HER-2 Group: Participant with Human epidermal growth factor (Her2/neu)-amplified tumor type (also positive for ER and PgR) who received 100 mg dasatinib BID.
- Participant CA180088-16-88002, ER and/or PgR Group: Participant with ER and PgR-amplified tumor type who received 100 mg dasatinib BID
- Participant CA180088-29-88085, ER and/or PgR Group: Participant with ER and PgR-amplified tumor type who received 70 mg dasatinib BID
Arm/Group | Participant CA180088-18-88009, HER-2 Group | Participant CA180088-16-88002, ER and/or PgR Group | Participant CA180088-29-88085, ER and/or PgR Group
Number analyzed (Participants) | 1 | 1 | 1
weeks | 31.14 | 18.14 | 8.29

9. Secondary Outcome: Number of Participants With Death, Adverse Events (AEs), and AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. AEs graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
Time Frame: Continuous assessment beginning at initiation of study drug until 30 days after the last dose of study drug
Population: All-Treated participants: All participants who received at least one dose of dasatinib.
Measure: Number; unit: participants
Groups:
- Dasatinib 70 mg: Dasatinib was administered orally at 70 mg BID, for a TDD of 140 mg.
- Dasatinib 100 mg: Dasatinib was administered orally at 100 mg BID, for a total daily dose (TDD) of 200 mg.
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 23 | 47
participants
  All Deaths | 6 | 6
  All AEs | 23 | 47
  AEs Leading to Discontinuation | 5 | 11

10. Secondary Outcome: Number of Participants With On-study CTCAE Version 3.0 Grade 3-4 Laboratory Abnormalities
Description: Normal ranges for laboratory abnormalities: granulocytes=1.5x10^3-8x10^3 mm^3 (range may have varied by institution); hemoglobin=12-16 g/dL; platelets=150-440x10^9c/L; partial thromboplastin time=27-37.1 seconds; alkaline phosphatase=38-126 U/L; alanine aminotransferase=15-48 U/L; aspartate aminotransferase=14-38 U/L; creatine=0.7-1.1 mg/dL; hypokalemia (potassium [K])=3.5-5mEq/L; hyponatremia (sodium [Na])=135-145 mEq/L; phosphorous=2.4-4.5 mg/dL; bilirubin=0-1.2. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening/disabling, Gr 5=Death.
Time Frame: Continuous assessment beginning at initiation of study drug until 30 days after the last dose of study drug
Population: All-Treated participants: All participants who received at least one dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 23 | 47
participants
  Granulocytes | 1 | 1
  Hemoglobin | 0 | 1
  Platelet Count | 0 | 1
  Partial Thromboplastin Time | 1 | 0
  Alkaline Phosphatase | 0 | 1
  Alanine Aminotransferase | 0 | 1
  Aspartate Aminotransferase | 1 | 3
  Creatinine | 1 | 0
  Hypokalemia | 1 | 0
  Hyponatremia | 0 | 1
  Phosphorous | 2 | 1
  Bilirubin | 0 | 1

11. Secondary Outcome: Number of Participants With Serious AEs (SAEs), Drug-related AEs, Drug-related SAEs, and Drug-Related Grade 3 AEs
Description: AEs and SAEs considered possibly, probably, or certainly related to study treatment, graded according to CTCAE Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death). SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: Continuous assessment beginning at initiation of study drug until 30 days after the last dose of study drug
Population: All-Treated participants: All participants who received at least one dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 23 | 47
participants
  Drug-related AEs | 22 | 44
  SAEs | 9 | 11
  Drug-related SAEs | 6 | 7
  Drug-related Grade 3 AEs | 9 | 15

12. Secondary Outcome: Number Of Participants With Notable Drug-related AEs
Description: Notable drug-related AEs for dasatinib include gastrointestinal symptoms (diarrhea, nausea, vomiting and abdominal pain), fatigue, lethargy, headache, rash, fever, pleural effusion, and dyspnea.
Time Frame: Continuous assessment beginning at initiation of study drug until 30 days after the last dose of study drug
Population: All-Treated participants: All participants who received at least one dose of dasatinib.
Measure: Number; unit: participants
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 23 | 47
participants
  Diarrhea | 10 | 22
  Nausea | 8 | 16
  Abdominal Pain | 2 | 11
  Fatigue | 3 | 17
  Rash | 8 | 11
  Pleural Effusion | 9 | 12
  Dyspnea | 9 | 10

13. Secondary Outcome: Pharmacokinetics (PK): Plasma Concentration of Dasatinib at Week 3
Description: Blood samples (3 mL) were used for measurement of dasatinib plasma concentration and metabolites.
Time Frame: PK assessment was performed at Week 3 visit (Day 15 ±4 days). Blood samples were obtained at Time = 0 hours, and at 1, 3 and 6 hours after each dose, and a trough sample was obtained immediately prior to any dose (~12 hours).
Population: Number of Participants Analyzed=All Treated Participants with samples for PK analysis, n=number of participants at specified time point with samples for PK analysis
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 17 | 14
ng/ml
  Time 0 hours (100 mg, n=16; 70 mg, n=13) | 10.82 (9.17) | 6.96 (2.90)
  Time 1 hour (100 mg, n=16; 70 mg, n=14) | 107.09 (64.55) | 77.21 (61.86)
  Time 3 hours (100 mg, n=17; 70 mg, n=14) | 58.01 (37.88) | 30.21 (18.42)
  Time 6 hours (100 mg, n=17; 70 mg, n=13) | 23.19 (15.20) | 12.64 (5.58)
  Time 12 hours (100 mg, n=16; 70 mg, n=9) | 11.88 (6.40) | 7.41 (5.08)

14. Secondary Outcome: PK: Plasma Concentration of Dasatinib at Week 7 or Week 9
Description: Blood samples (3 mL) were used for measurement of dasatinib plasma concentration and metabolites.
Time Frame: PK assessment was performed at Week 7 or 9 visit. Blood samples were obtained at Time = 0 hours, and at 1, 3 and 6 hours after each dose, and a trough sample was obtained immediately prior to any dose (~12 hours).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Dasatinib 50 mg: Dasatinib was administered orally at a starting dose of 70 mg BID. Dose adjustment was made according to tolerance, with reduction to 50 mg BID. Participants continued study treatment until PD or unacceptable toxicity. Dasatinib dose was adjusted so that drug-related toxicities were either Grade 0 - 1 or were Grade 2 toxicities that were adequately managed with outpatient therapy or deemed clinically acceptable.
Arm/Group | Dasatinib 100 mg | Dasatinib 70 mg | Dasatinib 50 mg
Number analyzed (Participants) | 5 | 9 | 1
ng/ml
  Time 0 hours (100 mg, n=5; 70 mg, n=7; 50 mg, n=1) | 9.49 (4.94) | 6.62 (3.54) | 6.06 (0.00)
  Time 1 hour (100 mg, n=5; 70 mg, n=8; 50 mg, n=1) | 131.09 (57.52) | 49.28 (37.97) | 4.75 (0.00)
  Time 3 hours (100 mg, n=5; 70 mg, n=9; 50 mg, n=1) | 55.26 (23.65) | 42.27 (21.94) | 35.74 (0.00)
  Time 6 hours (100 mg, n=5; 70 mg, n=8; 50 mg, n=1) | 23.58 (8.65) | 13.03 (3.34) | 35.91 (0.00)
  Time 12 hours (100 mg, n=4; 70 mg, n=6; 50 mg, n=1 | 10.52 (3.55) | 5.00 (2.26) | 9.02 (0.00)

15. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline In Plasma Level of Collagen Type IV at Week 3 in Participants With and Without DCR
Description: Collagen Type IV is a circulating marker related to the modulation of the vascular endothelial growth factor (VEGF)-pathway. An assay of Collagen Type IV in plasma was performed by ELISA.
Time Frame: At Baseline and Week 3 of treatment (Day 15 ±4 days)
Population: Number of Participants Analyzed=All Treated Participants with samples for PD analysis, n=number of participants at specified time point with samples for PD analysis
Measure: Mean (90% Confidence Interval); unit: percent change
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 29 | 19
percent change
  Participants with no DCR (n=27, n=16) | 32.07 [23.58 to 41.15] | 35.92 [25.72 to 46.94]
  Participants with DCR (n=2, n=3) | 22.01 [11.21 to 33.87] | 40.74 [10.81 to 78.75]
  All Participants (n=29, n=19) | 31.35 [23.46 to 39.76] | 36.67 [27.74 to 46.21]

16. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline In Plasma Level of Collagen Type IV at Week 5 in Participants With and Without DCR
Description: as for outcome 15
Time Frame: Week 5
Population: as for outcome 15
Measure: Mean (90% Confidence Interval); unit: percent change
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 23 | 15
percent change
  Participants with no DCR (n=20, n=12) | 45.37 [33.43 to 58.38] | 28.45 [-2.25 to 68.80]
  Participants with DCR (n=3, n=3) | 17.13 [-11.57 to 55.14] | 64.51 [34.18 to 101.68]
  All Participants (n=23, n=15) | 41.33 [30.41 to 53.18] | 34.97 [8.48 to 67.92]

17. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline In Plasma Level of VEGFR2 at Week 3 in Participants With and Without DCR
Description: VEGF-stimulated disruption of the cadherin-catenin complex leads to tumor cell invasion and metastasis. VEGFR2 plasma levels were assayed by ELISA as a marker of VEGF pathway modulation.
Time Frame: At Baseline and Week 3 of treatment (Day 15 ±4 days)
Population: as for outcome 15
Measure: Mean (90% Confidence Interval); unit: percent change
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 29 | 15
percent change
  Participants with no DCR (n=27, n=16) | 21.88 [15.98 to 28.08] | 23.61 [20.41 to 27.17]
  Participants with DCR (n=2, n=3) | 14.77 [6.25 to 23.97] | -5.03 [-55.67 to 103.43]
  All Participants (n=29, n=19) | 21.37 [15.88 to 27.13] | 18.57 [9.95 to 27.86]

18. Primary Outcome: Best Overall Response
Description: Response assessed using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR)=disappearance of all target and non-target lesions; Partial Response (PR)=≥30% decrease in sum of longest diameter (LD) of target lesions; SD=small changes not meeting above criteria; Progressive Disease (PD)=appearance of new lesion(s), ≥ 20% increase in the sum of the LD of target lesions, or progression of existing non-target lesions; Clinical Progression (cPD)=deterioration related to disease requiring treatment without radiographic PD.
Time Frame: From day of first treatment through Week 25 or at time of discontinuation from study treatment
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Her2/Neu-amplified Tumor, 70 mg Twice Daily (BID) Dasatinib | Her2/Neu-amplified Tumor, 100 mg BID | ER and/or PgR Positive Tumor, 70 mg BID Dasatinib | ER and/or PgR Positive Tumor, 100 mg BID Dasatinib
Number analyzed (Participants) | 15 | 9 | 31 | 14
participants
  Complete Response (CR) | 0 | 0 | 0 | 0
  Unconfirmed partial response | 0 | 0 | 1 | 0
  Partial Response (PR) | 0 | 1 | 1 | 1
  Stable Disease (SD) | 2 | 2 | 5 | 3
  Progressive Disease (PD) | 12 | 4 | 15 | 7
  Clinical Progression (cPD) | 0 | 1 | 3 | 1
  Discontinuation Due To Drug Toxicity (Tox) | 1 | 1 | 5 | 2
  No Reassessment -Reasons Other Than Tox/PD | 0 | 0 | 1 | 0

19. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline In Plasma Level of VEGFR2 at Week 5 in Participants With and Without DCR
Description: as for outcome 17
Time Frame: At Baseline and Week 5 of treatment
Population: as for outcome 15
Measure: Mean (90% Confidence Interval); unit: percent change
Arm/Group | Dasatinib 70 mg | Dasatinib 100 mg
Number analyzed (Participants) | 23 | 15
percent change
  Participants with no DCR (n=20, n=12) | 27.23 [22.53 to 32.10] | 26.36 [20.85 to 32.13]
  Participants with DCR (n=3, n=3) | 16.46 [8.27 to 25.27] | 37.25 [23.08 to 53.05]
  All Participants (n=23, n=15) | 25.77 [21.51 to 30.18] | 28.47 [23.48 to 33.66]

ADVERSE EVENTS:
Groups:
- Dasatinib: Dasatinib was administered orally at 70 mg BID (TDD=140 mg) or 100 mg BID (TDD=200 mg).
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 20/70
Other Adverse Events (participants affected / at risk) | 65/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=70)
WEIGHT INCREASED (Investigations) | 1
HEADACHE (Nervous system disorders) | 2
HEMIPARESIS (Nervous system disorders) | 1
BRAIN OEDEMA (Nervous system disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
PNEUMONIA (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
LOBAR PNEUMONIA (Infections and infestations) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1
FALL (Injury, poisoning and procedural complications) | 1
TOOTH INJURY (Injury, poisoning and procedural complications) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
FATIGUE (General disorders) | 2
PYREXIA (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=70)
LACRIMATION INCREASED (Eye disorders) | 4
WEIGHT DECREASED (Investigations) | 8
HAEMOGLOBIN DECREASED (Investigations) | 4
ALANINE AMINOTRANSFERASE (Investigations) | 5
ASPARTATE AMINOTRANSFERASE (Investigations) | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 10
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 12
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 6
PERICARDIAL EFFUSION (Cardiac disorders) | 7
INSOMNIA (Psychiatric disorders) | 4
HEADACHE (Nervous system disorders) | 28
DIZZINESS (Nervous system disorders) | 5
NAUSEA (Gastrointestinal disorders) | 26
VOMITING (Gastrointestinal disorders) | 17
DIARRHOEA (Gastrointestinal disorders) | 34
DYSPEPSIA (Gastrointestinal disorders) | 4
CONSTIPATION (Gastrointestinal disorders) | 7
ABDOMINAL PAIN (Gastrointestinal disorders) | 15
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 9
ANOREXIA (Metabolism and nutrition disorders) | 17
ANAEMIA (Blood and lymphatic system disorders) | 6
RASH (Skin and subcutaneous tissue disorders) | 19
ALOPECIA (Skin and subcutaneous tissue disorders) | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 11
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 24
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 19
CHILLS (General disorders) | 6
FATIGUE (General disorders) | 19
PYREXIA (General disorders) | 14
ASTHENIA (General disorders) | 24
CHEST PAIN (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.